CLINICAL TRIAL: NCT07291947
Title: Phase I/II Clinical Study of Personalized Ultra-fractionated Stereotactic Adaptive Radiotherapy (PULSAR) Combined With Immunotherapy and Chemotherapy in Patients With Cholangiocarcinoma
Brief Title: PULSAR Combined With Immunotherapy and Chemotherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wang Xin (Other)
Responsible Party: Sponsor-Investigator, Wang Xin, Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PULSAR-ICON
Record Dates: First submitted 2025-08-29; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cholangiocarcinoma
Keywords: locally advanced or metastatic cholangiocarcinoma; PULSAR; immunotherapy; chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Drug Therapy; DEAE-Dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PULSAR Combined with Immunotherapy and Chemotherapy (Experimental): PULSAR Combined with Immunotherapy and Chemotherapy
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection (QL1706); Radiation: PULSAR

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) — GC chemotherapy and Iparomlimab and Tuvonralimab Injection
  Other Names: chemotherapy
Radiation: PULSAR — Personalized Ultra-fractionated Stereotactic Adaptive Radiotherapy

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of PULSAR in combination with dual immune checkpoint inhibitors (PD-1 monoclonal antibody + CTLA-4 monoclonal antibody) and GC chemotherapy in patients with locally advanced or metastatic cholangiocarcinoma. The secondary objective of this study is to investigate the immunological impact of PULSAR combined with dual immune therapy (PD-1 monoclonal antibody + CTLA-4 monoclonal antibody) on the tumor microenvironment and systemic immune responses in cholangiocarcinoma patients.

DETAILED DESCRIPTION:
After confirmation of eligibility, enrolled patients will undergo radiation CT simulation and planning per standard of care. IV contrast will be administered with CT simulation at the treating physician's discretion though is not required.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent. The subject has fully understood and accepted the purpose, content, expected efficacy, mechanism of action, and risks of the study, and has signed the informed consent form.
2. Age 18-75 years, regardless of gender.
3. Histopathologically or cytologically confirmed locally advanced or metastatic cholangiocarcinoma.
4. At least one measurable lesion based on RECIST 1.1 criteria.
5. ECOG performance status score of 0-1.
6. Expected survival time ≥3 months.
7. Willing to comply with study procedures and able to undergo treatment (including radiotherapy, immunotherapy, chemotherapy) and follow-up.
8. No contraindications to the use of PD-1, PD-L1 inhibitors, gemcitabine, or cisplatin.
9. No contraindications to radiotherapy.
10. Organ function levels meet the following requirements: - Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; - Platelet (PLT) count ≥ 80 × 10⁹/L; - Hemoglobin (Hb) level ≥ 90 g/L; - Total bilirubin (TBil) level ≤ 1.5 times the upper limit of normal (ULN); - Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN; if liver metastases are present, ≤ 5 times ULN; - Serum creatinine ≤ 1.5 times ULN, or calculated creatinine clearance rate ≥ 50 ml/min; - International normalized ratio (INR) ≤ 1.5 times ULN, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN, unless the subject is receiving anticoagulant therapy. - Hepatitis B surface antigen (HBsAg) positive with peripheral blood hepatitis B virus DNA (HBV-DNA) titer ≤ 1 × 10³ copies/L; if HBsAg positive and peripheral blood HBV-DNA titer ≥ 1 × 10³ copies/L, subjects may be included if the investigator determines that the chronic hepatitis B is stable and poses no additional risk.
11. Women of childbearing potential must agree to use appropriate contraceptive measures during the study period. Additionally, a serum or urine pregnancy test performed within 24 hours prior to the initiation of chemotherapy must be negative.
12. Women must be non-lactating.

Exclusion Criteria:

1. Previously treated with anti-PD-1 or anti-PD-L1 antibodies.
2. Received any investigational drug treatment within 4 weeks prior to the first administration of the study drug.
3. Simultaneous participation in other clinical studies, unless it is an observational (non-interventional) clinical study or the follow-up phase of an interventional clinical study.
4. Previously received radiotherapy to the upper abdomen.
5. Uncontrolled severe diseases that the investigator considers may affect the subject's ability to receive study protocol treatment, such as severe cardiac disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infections, active peptic ulcers, etc.
6. Active known or suspected autoimmune diseases (including but not limited to uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilator treatment). Patients with hypothyroidism requiring hormone replacement therapy and those with skin conditions not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia) may be included.
7. Active tuberculosis infection. Patients with active pulmonary tuberculosis infection within the past year will be excluded, even if treated. Patients with a history of active pulmonary tuberculosis infection more than one year ago will also be excluded unless evidence is provided that they have undergone standard anti-tuberculosis treatment.
8. Patients requiring long-term systemic corticosteroid therapy (equivalent to >10 mg prednisone/day) or any other form of immunosuppressive therapy. Patients using inhaled or topical corticosteroids may be included.
9. Uncontrolled cardiac disease, such as: New York Heart Association (NYHA) Class II or higher heart failure; unstable angina; myocardial infarction within the past year; clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention. Additionally, dementia, altered mental status, or any psychiatric disorders that could impair the ability to understand, provide informed consent, or complete questionnaires.
10. History of allergy or hypersensitivity to any component of the treatment.
11. History of malignant tumors within the past 5 years, except for completely treated basal cell carcinoma or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, or ductal carcinoma in situ of the breast after radical surgery.
12. Previously received systemic therapy for cholangiocarcinoma.
13. Positive for hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies.
14. Active infection requiring systemic treatment.
15. Other conditions deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Safety of immunotherapy and chemotherapy combined with PULSAR radiation therapy | Baseline, every three weeks in the treatment period, 30 days and 3 months after treatment
  Evaluation of reported adverse events (AEs) and serious adverse events (SAEs), according to CTCAE v5.0.
  Evaluation of changes from Baseline during the Treatment and Follow-up periods

SECONDARY OUTCOMES:
immunological impact of immunotherapy and chemotherapy combined with PULSAR radiation therapy | Baseline, every three weeks in the treatment period, 30 days and 3 months after treatment
  Evaluation of immunological impact of PULSAR combined with dual immune therapy (PD-1 monoclonal antibody + CTLA-4 monoclonal antibody) on the tumor microenvironment and systemic immune responses in cholangiocarcinoma patients according to flow cytometry. Evaluation of changes from Baseline during the Treatment and Follow-up periodsTo investigate the

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided